CLINICAL TRIAL: NCT00562276
Title: Immediate Versus Delayed IUD Insertion Following Suction Aspiration Between 5 and 12 Weeks Gestation: a Randomized Trial
Brief Title: Immediate Versus Delayed Intrauterine Device (IUD) Insertion Following First Trimester Suction Aspiration Procedures
Acronym: PAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Paula Bednarek, Assistant Professor SM.OB/GYN Generalist Division, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OHSU FAMPLAN 2535
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Contraception
Keywords: IUD; insertion timing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Immediate IUD insertion following suction aspiration between 5 and 12 weeks gestation
  Interventions: Procedure: Immediate IUD insertion
- 2 (No Intervention): Delayed IUD insertion 2-6 weeks following suction aspiration between 5 and 12 weeks gestation

INTERVENTIONS:
Procedure: Immediate IUD insertion — Insertion of either Paraguard or Mirena IUD within minutes of completing suction aspiration procedure between 5 and 12 weeks gestation
  Arms: 1

SUMMARY:
The purpose of this multi-center clinical trial is to evaluate the safety and effectiveness of inserting an intrauterine device (IUD) immediately after a suction aspiration procedure compared to inserting the IUD 2-6 weeks after the procedure. This study will also evaluate how satisfied women are with the timing of their IUD placement. Subjects will be able to choose between the Paraguard IUD or the Mirena IUD.

The researchers hypothesize that:

1. the expulsion rates measured at 1, 3 and 6 months will be clinically equivalent with immediate insertion compared with delayed insertion,
2. satisfaction and tolerance of side effects will be higher with immediate IUD insertion compared with delayed insertion, and
3. overall IUD use/continuation rates measured at 1, 3 and 6 months will be higher with immediate IUD insertion compared with delayed insertion.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years or older
* Requesting suction aspiration for spontaneous or elective abortion
* Intrauterine pregnancy documented with ultrasound. For women with a gestational sac, the gestational age (EGA) must be ≥ 5 weeks 0 days but ≤ 12 weeks 0 days based on the following criteria:

  * If no embryonic pole present: EGA (days) = mean sac diameter (mm) + 30 (Mean sac diameter =[length+width+depth]/3)
  * If embryonic pole is present: EGA (days) determined by Hadlock scale for measured crown-rump length
* Desiring intrauterine contraception
* In general good health
* Willing and able to undergo informed consent
* Willing to comply with randomization and study follow-up schedule

Exclusion Criteria:

* Pelvic exam with evidence of active cervicitis or PID (eg. purulent discharge, adnexal mass, significant cervical or uterine tenderness)
* PID or sexually transmitted infection within the previous three months
* History of pelvic Actinomyces
* Unexplained vaginal bleeding
* Uterine anomaly (eg. bicornuate uterus)
* Leiomyomata that distort the uterine cavity
* Known or suspected complete molar pregnancy
* Current confirmed or possible ectopic pregnancy
* AIDS without treatment (individuals with HIV/AIDS who are clinically well are not excluded)
* Any prior surgical aspiration during this current pregnancy
* Use of osmotic dilators (eg. laminaria) or misoprostol for cervical preparation during the aspiration procedure
* Allergy to polyethylene
* Allergy to levonorgestrel (for levonorgestrel-containing IUS only)
* Allergy to copper (for copper T380A IUD only)
* Wilson's disease (for copper T380A IUD only)
* Current participation in another research study which would interfere with the conduct of this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
IUD expulsion | 1, 3 and 6 months after insertion

SECONDARY OUTCOMES:
IUD continuation | 1, 3 and 6 months after insertion

CONTACTS AND LOCATIONS:
Overall Officials: Paula H Bednarek, MD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - University of New Mexico, Albuquerque, New Mexico
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Bednarek PH, Creinin MD, Reeves MF, Cwiak C, Espey E, Jensen JT; Post-Aspiration IUD Randomization (PAIR) Study Trial Group. Prophylactic ibuprofen does not improve pain with IUD insertion: a randomized trial. Contraception. 2015 Mar;91(3):193-7. doi: 10.1016/j.contraception.2014.11.012. Epub 2014 Nov 25. PMID 25487172
- [Derived] Bednarek PH, Creinin MD, Reeves MF, Cwiak C, Espey E, Jensen JT; Post-Aspiration IUD Randomization (PAIR) Study Trial Group. Immediate versus delayed IUD insertion after uterine aspiration. N Engl J Med. 2011 Jun 9;364(23):2208-17. doi: 10.1056/NEJMoa1011600. PMID 21651392